CLINICAL TRIAL: NCT02434211
Title: Interventional Research in Schools - Second Part
Acronym: RISCOLAIRE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Laboratoire ACTé (Unknown); Education Nationale (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-03
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaire and Focus group (Experimental): The children complete the questionnaire to better know their knowledge and cancer individual conceptions. Then, they will be interviewed during one hour in groups for the pre-testing phase. And after, for the testing phase, they just complete the questionnaire.
  Interventions: Other: Questionnaire and focus group

INTERVENTIONS:
Other: Questionnaire and focus group

SUMMARY:
The main objective this project is the development of a measurement tool. This consists of construct and validate a questionnaire to conduct a quantitative assessment of knowledge and individual conceptions of cancer enrolled in CM1 and CM2 (9-11 years).

DETAILED DESCRIPTION:
* exper judges by DELPHI method for content validity
* pre-testing for appearence validity
* testing for construct validity

ELIGIBILITY:
Inclusion Criteria:

* children enrolled in classes CM1 and CM2 of the departments of Loire, Essonne, Rhone and Ain

Exclusion Criteria:

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 291 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Questionnaire validity | 1 hour